CLINICAL TRIAL: NCT04692051
Title: A Phase II Study for Nab-paclitaxel Plus Cisplatin vs Gemcitabine Plus Cispatin as First Line Chemotherapy in Advanced Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xianglin Yuan, Professor, Head of the cancer center, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-BTC-03
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Biliary Tract Cancer
Keywords: Nab-paclitaxel + Cisplatin
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-paclitaxel + Cisplatin (Experimental): Patients in this arm receive chemotherapy with Nab-paclitaxel plus Cisplatin
  Interventions: Drug: Nab-paclitaxel + Cisplatin
- Gemcitabine + Cisplatin (Active Comparator): Patients in this arm receive chemotherapy with Gemcitabine plus Cisplatin
  Interventions: Drug: Gemcitabine + Cisplatin

INTERVENTIONS:
Drug: Nab-paclitaxel + Cisplatin — Nab-paclitaxel 125mg/m2 IV on D1,8 plus Cisplatin 75mg/m2 IV on D1 , every 21 days.
  Arms: Nab-paclitaxel + Cisplatin
Drug: Gemcitabine + Cisplatin — Gemcitabine1000mg/m2 IV on D1,8 plus Cisplatin 75mg/m2 IV on D1 , every 21 days.
  Arms: Gemcitabine + Cisplatin

SUMMARY:
It is a trial to compare the efficacy and safety of Nab-paclitaxel plus Cisplatin vs Gemcitabine plus Cispatin as first line chemotherapy in advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years;
2. Diagnosis of unresectable or recurrent or metastatic biliary tract cancer (Ampulla of Vater, gallbladder, intra or extra-hepatic biliary ducts);
3. Adequate bone marrow, liver and kidney function: absdute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelet count (PLT) ≥75 x 10^9/L, hemoglobin (HB) ≥ 75 g/L, White blood cell(WBC) ≥ 3.0 x 10^9/L, no bleeding symptoms or bleeding tendency; Total bilirubin (TBIL) ≤ 3 x upper limit of normal range (ULN), alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤ 5 x upper limit of normal range (ULN); creatinine(Cr) ≤ 1.5 x upper limit of normal range(ULN) or creatinine clearance rate（CCR）≥ 45ml/min;
4. At least one measurable lesion;
5. Karnofsky Performance Status(KPS) ≥ 70;
6. Estimated life expectancy of at least 3 months;
7. Resolution of all acute clinical toxic effects of any prior treatment to grade ≤ 1, with the exception of alopecia;
8. Be able to understand and willingness to sign IRB-approved informed consent; (If the patient cannot sign the informed consent due to consciousness disorder, upper limbs paralysis or inability to write, the legal representative shall sign the informed consent on behalf of the patient).

Exclusion Criteria:

1. Ongoing uncontrolled infections, or have received systemic antibiotic therapy within 72 hours prior to registration;
2. Myeloproliferative disorder or any other hematopoietic function disorder;
3. Have an untreated second malignancy or brain metastasis;
4. Allergic to the chemotherapy drugs of this protocol;
5. Unable to cooperate due to neurologic diseases or psychiatric illness;
6. Pregnant or lactating female patients; Women of child-bearing age who refuse to accept contraceptive measures;
7. Have other significant medical illness, for example,active tuberculosis, active pneumonia, uncorrected electrolyte disturbance, uncontrolled tumor associated pain, uncontrolled hydrothorax or seroperitoneum and so on;
8. Patients need to receive other antitumor therapy at the same time;
9. Have received any other experimental treatment or participated in another interventional clinical trial within 30 days prior to registration;
10. Any other situation that the researcher considered patients are unsuitable for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years
  PFS is defined as time from the start of treatment to progression of disease or death.

SECONDARY OUTCOMES:
ORR | up to 3 years
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
OS | up to 3 years
  Overall survival is defined as time from the start of treatment until death due to any reason.
TTP | up to 3 years
  Time to progress is defined as time from randomized grouping to objective progression of tumors.
AEs | up to 3 years
  Adverse reactions refer to the occurrence and development of diseases in the process of using drugs according to normal usage and dosage to prevent, diagnose or treat diseases.Adverse reactions unrelated to the purpose of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yang X, Dai YH, Peng H, Zhang MS, Fu Q, Liu SF, Sun L, Zou YM, Xu HS, Qiu P, Qiu H, Huang Q, Cheng HH, Zhuang L. Nab-paclitaxel plus cisplatin versus gemcitabine plus cisplatin as first-line treatment in advanced biliary tract cancer: results of a multicentre, randomised, phase II trial. BMC Cancer. 2025 Aug 16;25(1):1321. doi: 10.1186/s12885-025-14581-3. PMID 40819029